CLINICAL TRIAL: NCT06513949
Title: Phase 2, Randomized, Double-Blind, Placebo-Controlled, Safety and Efficacy Study of Anti-CD14 Treatment With a Recombinant Chimeric Monoclonal Antibody (IC14) in Hospitalized Patients With Acute Respiratory Distress Syndrome
Brief Title: Anti-CD14 Treatment With IC14 in Hospitalized ARDS Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Implicit Bioscience (Industry)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARDS01
Record Dates: First submitted 2024-06-27; First posted 2024-07-22 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Acute Respiratory Distress Syndrome; Adult Respiratory Distress Syndrome; Acute Lung Injury; Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS)
Keywords: ARDS; IC14
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury | interventions — atibuclimab

STUDY DESIGN:
Intervention Model Description: Patients hospitalized with ARDS will be randomized to treatment with anti-CD14 monoclonal antibody, IC14, or placebo and evaluated for impact of treatment on severity of lung injury as measured by day 4 oxygenation index. Secondary objectives include determination of systemic and alveolar inflammatory responses; indices of oxygenation and illness severity; safety; and IC14 levels in bronchoalveolar lavage fluid and serum. Exploratory objectives include determining the effect of treatment on duration of mechanical ventilation, mortality, and feasibility of measuring presepsin, a CD14 pathway-specific biomarker at baseline using rapid testing
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical-appearing placebo prepared by research pharmacist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IC14 (atibuclimab) (Experimental): IC14 (atibuclimab) is a recombinant monoclonal antibody against human CD14
  Interventions: Biological: Atibuclimab
- Identical-appearing placebo (Placebo Comparator): Sterile normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Atibuclimab — monoclonal antibody against human CD14
  Other Names: IC14
  Arms: IC14 (atibuclimab)
Other: Placebo — Sterile normal saline for injection
  Arms: Identical-appearing placebo

SUMMARY:
Hospitalized patients with ARDS will be randomized to intravenous treatment with a monoclonal antibody against CD14, called IC14, or placebo. They will be followed for 28 days.

The primary outcome is the day 4 oxygenation index assessed as a continuous measure.

DETAILED DESCRIPTION:
This is a phase 2, randomized, double-blind, placebo-controlled, safety and efficacy study of anti-CD14 treatment with a recombinant chimeric monoclonal antibody (IC14) in hospitalized patients with Acute Respiratory Distress Syndrome (ARDS). CD14 is a key mediator in recognition of molecular markers of tissue damage (damage-associated molecular patterns, DAMPs) and infection (pathogen-associated molecular patterns, PAMPS).

The primary objective of the study is to determine the efficacy of IC14 in patients hospitalized with ARDS for reducing the severity of lung injury as measured by the day 4 Oxygenation Index (OI) assessed as a continuous measure (mean airway pressure x fraction of inspired oxygen [FiO2] x 100/partial pressure of oxygen [PaO2]). OI captures severity of hypoxemia and concurrent intensity of ventilatory support.

Secondary objectives include determining whether IC14 reduces the systemic and alveolar inflammatory response, and improves indices of oxygenation and illness severity. Exploratory endpoints include determining the effect of CD14 blockade on duration of mechanical ventilation and mortality in patients hospitalized with ARDS. Pharmacokinetic [PK]/Pharmacodynamic [PD] endpoints include determining day 4 IC14 levels in bronchoalveolar fluid (BALF) vs. serum, and determining the feasibility of measuring blood presepsin levels, a CD14-pathway specific biomarker for rapid assessment.

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if they meet all the following criteria:

1. Adult patients (18+) on mechanical ventilations with acute respiratory distress syndrome (ARDS) by Berlin Criteria (≤48 hours)

   1. P:F ratio < 300
   2. Positive end-expiratory pressure (PEEP) ≥5 cm H2O
   3. Bilateral opacities on chest x-ray or chest computerized tomography (CT)-- not fully explained by effusions, lobar/lung collapse, or nodules
   4. Respiratory failure not fully explained by cardiac failure or fluid overload
   5. Within 1 week of known clinical insult or new or worsening respiratory symptoms

   i. Common Risk Factors for ARDS: Pneumonia, aspiration, inhalation injury, pulmonary contusion, pulmonary vasculitis, drowning, non-pulmonary sepsis, major trauma, pancreatitis, severe burns, non-cardiogenic shock, drug overdose, multiple transfusions
2. Patient or Legal authorized representative able to understand and give written informed consent

Exclusion Criteria:

An individual fulfilling any of the following criteria should be excluded from enrollment in the study:

1. Significant pre-existing organ dysfunction prior to hospitalization

   1. Lung: Currently receiving home oxygen therapy as documented in medical record
   2. Heart: Pre-existing congestive heart failure defined as an ejection fraction <20% as documented in the medical record
   3. Renal: End-stage renal disease requiring renal replacement therapy or estimated glomerular filtration rate (eGFR) <30 mL/min.
   4. Liver: Severe chronic liver disease defined as Child-Pugh Class C or hepatic transaminases >5 times upper limit of normal
   5. Hematologic: Baseline platelet count <50,000/mm3
2. Presence of co-existing infection, including, but not limited to:

   1. HIV infection not virally suppressed and with pre-hospitalization CD4 counts ≤ 500 cell/mm3
   2. Active tuberculosis or a history of inadequately treated tuberculosis
   3. Active hepatitis B or hepatitis C viral infection
3. Current treatment, or treatment within 30 days or five half-lives (whichever is longer) with etanercept (Enbrel®), infliximab (Remicade®), adalimumab (Humira®), certolizumab (Cimzia®), golimumab (Simponi®), anakinra (Kineret®), rilonacept (Arcalyst®), tocilizumab (Actemra®), sarilumab (Kevzara®), siltuximab (Sylvant®), or other potent immunosuppressant or immunomodulatory drugs or treatments
4. Receiving comfort measures only
5. Requiring >2 vasopressors
6. Pregnant
7. Prisoners
8. History of hypersensitivity or idiosyncratic reaction to IC14
9. Women who are currently breastfeeding
10. Bronchoscopy safety exclusions

    1. P:F <100 on 100% FiO2
    2. Mean pulmonary artery pressure > 55 mmHg
    3. Marked cardiovascular instability (Mean arterial pressure <55 mmHg with vasopressor support)
    4. Intracranial pressure ≥20 mmHg
    5. Acute ischemic heart disease (unstable angina or ST-elevation myocardial infarction or Type 1 non-ST-elevation myocardial infarction)
    6. Supported on extracorporeal membrane oxygenation
    7. Endotracheal tube <6.5 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Day 4 Oxygenation Index | Day 1 through Day 4
  (mean airway pressure x fraction of inspired oxygen [FiO2] x100)/ partial pressure of oxygen [PaO2]

SECONDARY OUTCOMES:
Biomarkers of injury and inflammation measured in bronchoalveolar lavage fluid | Day 4
  Interleukin(IL)-6
Biomarkers of injury and inflammation measured in plasma | Day 4
  Interleukin(IL)-6
Oxygenation index | Days 7 and 14
  (mean airway pressure x FiO2 x100)/PaO2
Oxygen saturation index | Days 4, 7, and 14
  (mean airway pressure x FiO2 x100)/peripheral oxygen saturation [SpO2]
P:F ratio | Days 4, 7, and 14
  Ratio of partial pressure of arterial oxygen (P) to fraction of inspired oxygen (F)
S:F ratio | Days 4, 7, and 14
  Ratio of the arterial oxygen saturation (S) to fraction of inspired oxygen (F)
Sequential Organ Failure Assessment (SOFA) Score (range 0 [best] to 24 [worst]) | Days 4, 7, and 14
  Disease severity scale
Time to blood presepsin level | Days 0-4
  Time from study consent to measurement completion of blood presepsin level via the PATHFASTTM instrument
Cumulative incidence of run failures | Days 0-1
  Defined as not completing presepsin measurement between consent and infusion of study drug
Cumulative incidence of protocol-specified exempt serious events | Days 1-28
  protocol-specified exempt serious events
Cumulative incidence of grade 3 and 4 clinical and laboratory adverse events | Days 1-28
  Common Toxicity Criteria for Adverse Events version 5.0
Cumulative incidence of serious adverse events | Days 1-28
  Serious adverse events standard definition
Cumulative incidence of adverse events of special interest | Days 1-28
  Adverse events of special interest for test article and bronchoalveolar lavage

OTHER OUTCOMES:
Ventilator-free Days | Days 1-28
  Days alive and free of invasive mechanical ventilation
Mortality | Day 1-28
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Linzee Mabrey, MD, MsC, Principal Investigator — Unversity of Washington
Locations (2):
- United States (2):
  - Harborview Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No